CLINICAL TRIAL: NCT06428214
Title: A Post-market, Open-label, 3-Armed, Parallel Group, Multicenter Study to Evaluate Aesthetic Improvement and Safety of Restylane Shaype for Temporary Augmentation of the Chin Region Alone or in Combination With Restylane Defyne and Restylane Lyft Lidocaine Treatment in the Lower Face and Midface
Brief Title: A Restylane Treatment Algorithm Approach for Participants With Appearance of Insufficient Bone Structure in the Lower Face Alone or in Combination With Facial Soft Tissue Deficiencies
Acronym: ARTIST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05DF2307
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2024-05

CONDITIONS: Chin Augmentation
Keywords: lower face; Mid face

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Restylane Shaype (Experimental): Participants will receive Restylane Shaype in the chin area only.
  Interventions: Device: Restylane Shaype
- Restylane Shaype with Restylane Defyne (Other): Participants will receive Restylane Shaype in the chin area and Restylane Defyne in the marionette line areas laterally to the chin.
  Interventions: Device: Restylane Shaype; Device: Restylane Defyne
- Restylane Shaype with Restylane Defyne and Restylane Lyft Lidocaine (Other): Participants will receive Restylane Shaype in the chin area and Restylane Defyne in the marionette line areas laterally to the chin. Participants in this group will be treated with Restylane Lyft lidocaine in the midface, nasolabial folds (NLF) and /or jawline.
  Interventions: Device: Restylane Shaype; Device: Restylane Defyne; Device: Restylane Lyft lidocaine

INTERVENTIONS:
Device: Restylane Shaype — Injection
Device: Restylane Defyne — Injection
  Arms: Restylane Shaype with Restylane Defyne; Restylane Shaype with Restylane Defyne and Restylane Lyft Lidocaine
Device: Restylane Lyft lidocaine — Injection
  Arms: Restylane Shaype with Restylane Defyne and Restylane Lyft Lidocaine

SUMMARY:
The study's main purpose is to evaluate the overall aesthetic improvement of the treated areas by treatment group, as assessed by the Investigator.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing to comply with the requirements of the study including being photographed, following post-treatment care instructions, attending all study visits and providing a signed written informed consent.
* Males or non-pregnant, non-breastfeeding females, over the age of 18.
* Intent to receive treatment for temporary augmentation in the chin region.

Exclusion Criteria:

* Known/previous allergy or hypersensitivity to any injectable hyaluronic acid (HA) gel or to gram positive bacterial proteins and/or local anesthetics, e.g., lidocaine or other amide-type anesthetics
* Previous or present multiple allergies or severe allergies, such as manifested by anaphylaxis or angioedema, or family history of these conditions.
* Previous facial surgery (including facial aesthetic surgery and liposuction), below the level of the horizontal line from the lower orbital rim.
* Any previous aesthetic procedures or implants.
* Use of concomitant medication that have the potential to prolong bleeding times such as anticoagulants or inhibitors of platelet aggregation.
* Participation in any other interventional clinical study within 30 days (about 4 and a half weeks) before baseline.
* Women who are pregnant or breast feeding, or women of childbearing potential who are not practicing adequate contraception or planning to become pregnant during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2024-05-13 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2024-09-24 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Rated "Improved" or "Much Improved" or "Very Much Improved" as Assessed by Investigator Using the Global Aesthetic Improvement Scale (GAIS) at Week 8 | At week 8

SECONDARY OUTCOMES:
Percentage of Participants Rated "Improved" or "Much Improved" or "Very Much Improved" as Assessed by Investigator Using the GAIS at Week 4 | At week 4
Percentage of Participants Rated "Improved" or "Much Improved" or "Very Much Improved" as Assessed by the Participant Using the GAIS at week 4 and 8 | At weeks 4 and 8
Percentage of Participants Reporting "Agree" or "Strongly Agree", "Satisfied" or "Very satisfied" as per Participant Satisfaction Questionnaire at Week 8 | At week 8
Percentage of Participants in Each Response Category for Every Question in the Participant Satisfaction Questionnaire at Week 8 | At week 8
Percentage of Investigators Reporting "Agree" or "Strongly agree" as per Investigator Satisfaction Questionnaire at Week 8 | At week 8
Percentage of Participants in Each Response Category for Every Question in the Investigator Satisfaction Questionnaire at Week 8 | At week 8

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Galderma Investigational Site # 8754, Vancouver, British Columbia
  - Galderma Investigational Site 8379, Burlington, Ontario
  - Galderma Investigational Site 8690, Westmount, Quebec